CLINICAL TRIAL: NCT05435573
Title: Coload Effect on Cardiac Output Measurement Using Transthoracic Echocardiography in Preeclamptic Patients Undergoing Cesarean Delivery
Brief Title: Cardiac Output in Preeclamptic
Acronym: Coload
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, maha abou-zeid, Assistant Professor of Anesthesia and Surgical Intensive Care, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECHO
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Echocardiography
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated via sealed opaque envelops into 2 groups of 17 patients each; crystalloid group and group crystalloid-colloid group
Who Masked: Participant, Investigator
Masking Description: All the fluids were prepared according to the group by an anesthetist who will not be involved in data collection. All the bottles were wrapped by opaque cover.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid group (Active Comparator): The patients will receive 1000 mL of ringer's acetate solution (250 mL over 5 minutes starting immediately after intrathecal injection using a pressurizer then 500 mL over 55 minutes then 250 mL over 60 minutes).
  Interventions: Drug: 1000 mL of ringer's acetate solution
- Crystalloid-colloid group (Active Comparator): Patients will receive 250 mL 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride starting immediately after intrathecal injection then 500 mL of ringer's acetate solution then 250 mL of hydroxyethyl starch
  Interventions: Drug: 250 mL 6% hydroxyethyl starch (Voluven) then 500 mL of ringer's acetate solution then 250 mL of 6% hydroxyethyl starch (Voluven)

INTERVENTIONS:
Drug: 1000 mL of ringer's acetate solution — 1000 mL of ringer's acetate solution
  Arms: Crystalloid group
Drug: 250 mL 6% hydroxyethyl starch (Voluven) then 500 mL of ringer's acetate solution then 250 mL of 6% hydroxyethyl starch (Voluven) — 500 mL 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride plus 500 mL of ringer's acetate solution
  Arms: Crystalloid-colloid group

SUMMARY:
There is high incidence of hypertensive disorders during pregnancy.The maternal cardiovascular system had significant changes during pregnancy. The colloid oncotic pressure is decreased during preeclampsia.

DETAILED DESCRIPTION:
Transthoracic echocardiography considered an accurate non-invasive device and has validity for measuring cardiac functions in pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pre-eclampsia
* Age 18-45 years.
* Singleton pregnancy scheduled for elective CS delivery under spinal anesthesia.
* American Society of Anesthesiologists (ASA Ⅱ, Ⅲ).

Exclusion Criteria:

* Body mass index < 18 or ≥40 kg/m²
* Women presenting in labor
* Current administration of vasoactive drugs including salbutamol and thyroxin.
* Diabetes mellitus.
* Hemoglobin <10 g/dl.
* Cardiovascular, cerebrovascular, or renal disease
* Increased serum creatinine level ≥1.1 mg/dL.
* Contraindications to spinal anesthesia:(increased intracranial pressure, coagulopathy, or local skin infection)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Singleton pregnant preeclampsia scheduled for elective cesarean section delivery under spinal anesthesia
Enrollment: 34 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measurement | 1 hour from the spinal anesthesia
  1 hour post spinal anesthesia after administration of 1000 mL fluid using Transthoracic Echocardiography

SECONDARY OUTCOMES:
Cardiac output measurement | 5 minutes after the spinal anesthesia, after delivery of the fetus and 2 hours post spinal anesthesia
  at baseline ,5 minutes after spinal anesthesia, after delivery of the fetus and 2 hours post spinal anesthesia
Left ventricular end diastolic volume (LVEDV) measurement | 1 hour from the spinal anesthesia
  milliliter
Urine output volume | 1hour and 2 hours post spinal anesthesia
  milliliters
Heart rate (HR) | basal (preoperative), intraoperative each 10 minutes and postoperatively every hour during first 6 hours
  beats per minute
Mean Blood pressure | basal (preoperative), intraoperative each 10 minutes and postoperatively every hour during first 6 hours
  mmHg

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University-Emergency hospital-ICU, Al Mansurah, Egypt